CLINICAL TRIAL: NCT00723528
Title: A Placebo-Controlled Double-Blind Comparative Study of CNTO1275 in Patients With Plaque Type Psoriasis
Brief Title: An Efficacy and Safety Study of Ustekinumab (CNTO 1275) in Participants With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015166; JNS009-JPN-02
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Psoriasis
Keywords: Psoriasis; Ustekinumab; CNTO 1275
MeSH Terms: conditions — Psoriasis | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (CP) (Placebo Comparator): Placebo 0.5 ml and 1.0 ml will be administered subcutaneously (SC) on Weeks 0 and 4 respectively during the controlled period (Weeks 0-12).
  Interventions: Drug: Placebo (CP)
- Ustekinumab 45 mg (CP) (Active Comparator): Ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) will be administered SC on Weeks 0 and 4 during controlled period (Weeks 0-12).
  Interventions: Drug: Ustekinumab 45 mg (CP)
- Ustekinumab 90 mg (CP) (Active Comparator): Ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) will be administered SC on Weeks 0 and 4 during controlled period (Weeks 0-12).
  Interventions: Drug: Ustekinumab 90 mg (CP)
- Placebo A (After CP) (Placebo Comparator): After the controlled period (that is [i.e.], during the active drug treatment period [Weeks 12-64]), the placebo group will be randomized into 2 groups, including Placebo A, in which ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) will be administered SC at Weeks 12, 16, 28, 40, and 52.
  Interventions: Drug: Placebo A (After CP)
- Placebo B (After CP) (Placebo Comparator): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), the placebo group will be randomized into 2 groups, including Placebo B, in which ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) will be administered SC at Weeks 12, 16, 28, 40, and 52.
  Interventions: Drug: Placebo B (After CP)
- Ustekinumab 45 mg (After CP) (Active Comparator): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 45 mg group will receive placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) SC at Weeks 16, 28, 40 and 52.
  Interventions: Drug: Ustekinumab 45 mg (After CP)
- Ustekinumab 90 mg (After CP) (Active Comparator): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 90 mg group will receive placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) SC at Weeks 16, 28, 40 and 52.
  Interventions: Drug: Ustekinumab 90 mg (After CP)

INTERVENTIONS:
Drug: Placebo (CP) — Placebo 0.5 ml and 1.0 ml will be administered subcutaneously (SC) on Weeks 0 and 4 respectively during the controlled period (Weeks 0-12).
  Arms: Placebo (CP)
Drug: Ustekinumab 45 mg (CP) — Ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) will be administered SC on Weeks 0 and 4 during controlled period (Weeks 0-12).
  Arms: Ustekinumab 45 mg (CP)
Drug: Ustekinumab 90 mg (CP) — Ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) will be administered SC on Weeks 0 and 4 during controlled period (Weeks 0-12).
  Arms: Ustekinumab 90 mg (CP)
Drug: Placebo A (After CP) — After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), the placebo group will be randomized into 2 groups, including Placebo A, in which ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) will be administered SC at Weeks 12, 16, 28, 40, and 52.
  Arms: Placebo A (After CP)
Drug: Placebo B (After CP) — After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), the placebo group will be randomized into 2 groups, including Placebo B, in which ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) will be administered SC at Weeks 12, 16, 28, 40, and 52.
  Arms: Placebo B (After CP)
Drug: Ustekinumab 45 mg (After CP) — After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 45 mg group will receive placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) SC at Weeks 16, 28, 40 and 52.
  Arms: Ustekinumab 45 mg (After CP)
Drug: Ustekinumab 90 mg (After CP) — After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 90 mg group will receive placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) SC at Weeks 16, 28, 40 and 52.
  Arms: Ustekinumab 90 mg (After CP)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ustekinumab (CNTO 1275) compared with placebo in participants with moderate to severe plaque type psoriasis.

DETAILED DESCRIPTION:
This is a multicenter (involving more than 1 study center), randomized (study medication assigned by chance), double-blind (neither the invesitigator nor the participant knows the identity of the study medication), placebo- controlled (1 of the study medications is inactive), parallel-group comparative study (different groups of participants will receive different treatments at the same time). The total duration of the study will be 78 weeks which will be comprised of: a screening period (6 weeks); an efficacy assessment period (64 weeks [with a total of 7 treatments at Weeks 0, 4, 12, 16, 28, 40, and 52]) and a follow-up assessment period (8 weeks). The efficacy assessment period will further include: a placebo-controlled treatment period (Weeks 0-12) and an active drug treatment period (Weeks 12-64). During the placebo-controlled treatment period, participants will receive ustekinumab (45 mg or 90 mg) subcutaneously (SC-into the muscles) or placebo SC. During the active drug treatment period, participants will continue treatment with 45 mg or 90 mg SC as assigned during the placebo-controlled treatment period; however, participants in the placebo group will be divided into 2 groups and will receive ustekinumab 45 mg (Placebo A) or 90 mg (Placebo B) SC. Efficacy will be evaluated primarily by analysis of psoriasis area and severity index (PASI) score. Participant safety will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with psoriasis (psoriasis vulgaris and psoriatic arthritis) at least 6 months before registration
* Participants with plaque type psoriasis covering at least 10 percent of total body surface area at the time of informed consent and at registration
* Participants with a PASI score of greater than or equal to 12 at the time of informed consent and at registration
* Female participants of childbearing potential or males, whose partner can be pregnant, must agree that he/she will continuously take an appropriate contraceptive measure for 1 year from the day of informed consent to termination of the final investigational treatment; in the case of childbearing potential females, pregnancy test at screening must be negative
* Participants must agree not to receive Bacillus Calmette-Guérin (BCG) vaccination and live vaccine inoculation for 1 year after final treatment with the investigational product

Exclusion Criteria:

* Participants with guttate psoriasis, erythrodermic psoriasis, or pustular psoriasis
* Participants with a medical history of tuberculosis infection or suspected tuberculosis infection
* Participants with present or past history of chronic or recurrent infection (e.g., chronic or recurrent urinary tract infection or respiratory infection)
* Participants with a current serious infection (e.g., sepsis, hepatitis, pneumonia, or pyelonephritis) or those who experienced a serious infection within the 2 month period before registration and including participants who received intravenous administration of antibiotics or antiviral agents within the 2 month period before registration
* Participants with a current or past history of malignant tumors (except for basal cell carcinoma, intraepidermal squamous cell carcinoma in the skin and uterine cervical squamous cell carcinoma, whose treatment was completed and no sign suggesting a recurrence has been observed, and squamous cell carcinoma in the skin whose treatment was completed and no sign suggesting a recurrence has been observed in the past 5 years)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (27):
- Japan (27):
  - Asahikawa
  - Chitose
  - Chūō
  - Fukuoka
  - Fushimi
  - Isehara
  - Kanazawa
  - Kurume
  - Kyoto
  - Maebashi
  - Minato
  - Morioka
  - Nagasaki
  - Nagoya
  - Nankoku
  - Nishinomiya
  - Osaka
  - Ōsaka-sayama
  - Sagamihara
  - Sapporo
  - Sendai
  - Shigenobu N/A
  - Shimotsuke
  - Shinjuku
  - Suita
  - Tokyo
  - Tsu

REFERENCES:
- See also: Week 28 data cut-off Clinical Study Report for a Placebo-Controlled Double-Blind Study of CNTO 1275 in Subjects with Plaque Psoriasis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=425&filename=CR015166_w28CSR.pdf
- See also: |Final Clinical Study Report for A Placebo-Controlled Double-Blind Study of CNTO 1275 in Subjects with Plaque Psoriasi — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=425&filename=CR015166_finalCSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (CP): Placebo 0.5 ml and 1.0 ml was administered subcutaneously (SC) on Weeks 0 and 4 respectively during the controlled period (Weeks 0-12).
- Ustekinumab 45 mg (CP): Ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) was administered SC on Weeks 0 and 4 during the controlled period (Weeks 0-12).
- Ustekinumab 90 mg (CP): Ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) was administered SC on Weeks 0 and 4 during the controlled period (Weeks 0-12).
- Placebo A (After CP): After the controlled period (that is [i.e.], during the active drug treatment period [Weeks 12-64]), the placebo group was randomized into 2 groups, including Placebo A, in which ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) was administered SC at Weeks 12, 16, 28, 40, and 52. Participants were then followed until Week 72.
- Placebo B (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), the placebo group was randomized into 2 groups, including Placebo B, in which ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) was administered SC at Weeks 12, 16, 28, 40, and 52. Participants were then followed until Week 72.
- Ustekinumab 45 mg (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 45 mg group received placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) SC at Weeks 16, 28, 40 and 52. Participants were then followed until Week 72.
- Ustekinumab 90 mg (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 90 mg group received placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) SC at Weeks 16, 28, 40 and 52. Participants were then followed until Week 72.
Period: Period 1: Controlled Period (CP)
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 32 | 64 | 62 | 0 | 0 | 0 | 0
Completed | 28 | 64 | 58 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 4 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Onset of Tuberculosis Infection | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal due to worsened symptoms | 2 | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 2: After Controlled Period
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Started | 0 | 0 | 0 | 15 | 13 | 64 | 58
Completed | 0 | 0 | 0 | 14 | 11 | 58 | 54
Not Completed | 0 | 0 | 0 | 1 | 2 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Onset of tuberculosis infection | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Use of prohibited concomitant medication | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal due to worsened symptoms | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Total
Number analyzed (Participants) | 31 | 64 | 62 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (12.7) | 46.6 (12.5) | 46.8 (12.8) | 47.0 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 15 | 31
  Male | 26 | 53 | 47 | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Greater Than or Equal to 75 Percent (%) Improvement in Psoriasis Area and Severity Index (PASI) Score
Description: Percentage of participants with >=75% improvement in PASI score at Week 12 from Baseline was reported. PASI is a widely used tool for the measurement of severity of psoriasis. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) to 72 (worst). Baseline visit refers to Week 0.
Time Frame: Week 12
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP)
Number analyzed (Participants) | 31 | 64 | 62
Percentage of participants | 6.5 | 59.4 | 67.7
Statistical Analysis 1: Comparison: Ustekinumab 45 mg (CP) vs Ustekinumab 90 mg (CP); Test type: Superiority or Other; p < 0.0001, Fisher Exact — Fisher's exact test (using Holm's method)

2. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a self-administered 10-item questionnaire that is used to assess 6 different aspects of quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Scores range from 0 (no impairment in quality of life) to 30 (most impairment in quality of life).
Time Frame: Week 12
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP)
Number analyzed (Participants) | 31 | 62 | 61
Units on scale | -0.3 (5.25) | -8.0 (6.45) | -7.4 (6.52)
Statistical Analysis 1: Comparison: Ustekinumab 45 mg (CP) vs Ustekinumab 90 mg (CP); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — 2-sample t-test (using Holm's method)

3. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: PASI is a widely used tool for the measurement of severity of psoriasis. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Time Frame: Week 64
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication. Here,'N' signifies the participants evaluated for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Placebo B (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), the placebo group was randomized into 2 groups, including Placebo B, in which ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) was administered SC at Weeks 12, 16, 28, 40, and 52.
- Ustekinumab 45 mg (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 45 mg group received placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 45 mg (0.5 ml) and placebo (1.0 ml) SC at Weeks 16, 28, 40 and 52.
- Ustekinumab 90 mg (After CP): After the controlled period (i.e., during the active drug treatment period [Weeks 12-64]), participants in the ustekinumab 90 mg group received placebo (0.5 ml and 1.0 ml) SC at Week 12 followed by ustekinumab 90 mg (1.0 ml) and placebo (0.5 ml) SC at Weeks 16, 28, 40 and 52.
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 14 | 60 | 56
Units on a scale | 10.83 (16.149) | 8.29 (9.975) | 6.60 (9.060) | 4.94 (7.493)

4. Secondary Outcome: Percentage of Treatment Response Based on Psoriasis Area and Severity Index (PASI) Score
Description: PASI is a widely used tool for the measurement of severity of psoriasis. The combination of redness, scaling, and thickness, as well as overall body involvement determine the PASI score. The scale ranges from 0 (best) to 72 (worst). Percentage of Treatment Response= (Baseline PASI score-PASI score after treatment)/Baseline PASI score x 100. Baseline visit refers to Week 0.
Time Frame: Week 64
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of treatment response
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 14 | 60 | 56
Percentage of treatment response | 70.78 (38.816) | 63.07 (43.608) | 78.86 (25.910) | 82.36 (26.798)

5. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (>=) 50 Percent (%), 90%, and Equal to 100% of Treatment Response Based on PASI Score
Description: as for outcome 4
Time Frame: Week 64
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication. Here, 'N' signifies the participants evaluated for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 14 | 60 | 56
Percentage of participants
  >= 50% Treatment Response | 80 | 71.4 | 91.7 | 89.3
  >= 90% Treatment Response | 60 | 50 | 50 | 55.4
  100% Treatment Response | 13.3 | 21.4 | 18.3 | 17.9

6. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Week 28, 40, 52 and 64
Description: as for outcome 2
Time Frame: Week 28, 40, 52 and 64
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication. Here,'N' signifies the participants evaluated for this measure and 'n' signifies the participants evaluated for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 15 | 64 | 59
Unit on scale
  Change at Week 28 (n=15,15,64,59) | -6.4 (6.74) | -6.2 (6.14) | -7.5 (6.46) | -7.6 (6.59)
  Change at Week 40 (n=15,15,61,56) | -6.5 (6.46) | -6.5 (6.08) | -7.7 (6.98) | -7.9 (6.62)
  Change at Week 52 (n=15,14,60,57) | -6.3 (5.92) | -5.5 (6.60) | -7.3 (7.01) | -7.8 (6.96)
  Change at Week 64 (n=15,14,60,56) | -5.8 (6.05) | -5.7 (6.96) | -7.4 (6.92) | -7.9 (6.43)

7. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) at Week 12, 28, 40, 52 and 64
Description: The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: (1) physical component summary (PCS)=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary (MCS)=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both sub scores and summary scores. For sub scores and summary scores: 0=worst score and 100=best score.
Time Frame: Week 12, 28, 40, 52 and 64
Population: The full analysis set (FAS) population included all the randomly assigned participants with efficacy data who fulfilled the eligibility criteria and received study medication. Here, 'N' signifies the participants evaluated for this measure and 'n' signifies the participants evaluated for this measure at a particular time point.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 16 | 64 | 61
Unit on scale
  Change at Week 12: PCS(n=15,16,62,61) | -.88 (11.141) | -1.03 (8.328) | 7.76 (14.536) | 5.14 (12.036)
  Change at Week 12: MCS(n=15,16,62,61) | 1.16 (5.263) | 2.84 (7.994) | 5.28 (9.797) | 5.77 (10.450)
  Change at Week 28: PCS(n=15,15,64,59) | 2.22 (15.064) | 6.42 (16.113) | 8.54 (14.538) | 6.23 (11.721)
  Change at Week 28: MCS(n=15,15,64,59) | 6.19 (7.069) | 3.22 (6.621) | 6.84 (10.086) | 7.24 (11.932)
  Change at Week 40: PCS(n=15,15,61,57) | 2.12 (19.683) | 6.18 (15.914) | 8.95 (15.476) | 3.58 (16.339)
  Change at Week 40: MCS(n=15,15,61,57) | 4.90 (5.453) | 5.27 (11.303) | 6.61 (9.674) | 8.34 (10.415)
  Change at Week 52: PCS(n=15,14,60,56) | 4.03 (16.426) | 6.58 (16.496) | 8.33 (16.365) | 6.19 (13.608)
  Change at Week 52: MCS(n=15,14,60,56) | 4.44 (5.198) | 5.93 (9.755) | 5 (10.386) | 7.69 (8.998)
  Change at Week 64: PCS(n=15,14,60,56) | 3.79 (15.519) | 6.10 (16.164) | 8.27 (15.468) | 6.70 (12.990)
  Change at Week 64: MCS(n=15,14,60,56) | 4.67 (5.362) | 5.21 (7.958) | 5.11 (10.504) | 6.89 (9.433)

8. Secondary Outcome: Change From Baseline in Psoriasis Disability Index (PDI) Score at Week 12, 28, 40, 52 and 64
Description: The PDI questionnaire consists of 15 questions relating to the impact of psoriasis in terms of daily activities, work or school, personal relationships, leisure, and treatment. Each question is scored on a scale of 0 (no impact) to 3 (greatest impact). The PDI is calculated by summing the scores of the questions resulting in a maximum score of 45 (greatest impact) and a minimum score of 0 (no impact).
Time Frame: Week 12, 28, 40, 52 and 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 16 | 64 | 61
Unit on scale
  Change at Week 12 (n=15,16,62,61) | 0.1 (3.70) | 0.1 (4.76) | -8.6 (9.63) | -12.0 (11.80)
  Change at Week 28 (n=15,15,64,59) | -10.0 (9.52) | -8.1 (8.90) | -10.8 (9.45) | -13.2 (10.75)
  Change at Week 40 (n=15,15,61,57) | -9.4 (9.07) | -8.5 (9.67) | -11.3 (9.92) | -14.0 (10.53)
  Change at Week 52 (n=15,14,60,56) | -10.4 (8.60) | -6.5 (10.86) | -10.6 (9.06) | -14.5 (10.64)
  Change at Week 64 (n=15,14,60,56) | -10.6 (9.12) | -7.6 (10.10) | -10.7 (9.71) | -14.3 (10.17)

9. Secondary Outcome: Treatment Response Based on Nail Psoriasis Severity Index (NAPSI) Score
Description: The NAPSI score is used to evaluate the severity of nail bed psoriasis and nail matrix psoriasis. The nail is divided with into quadrants and given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of any of the features of nail psoriasis in that quadrant. Each nail is evaluated, and the sum of all the nails is the total NAPSI score. The sum of the scores from all nails ranges from 0 (no psoriasis) to 80 (psoriasis present in all 4 quadrants of all 10 nails).
Time Frame: Week 12, 28, 40,52 and 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 9 | 8 | 44 | 40
Unit on scale
  NAPSI Score at Week 12 (n=9,8,43,40) | 11.1 (33.33) | 6.3 (17.68) | 7.7 (95.14) | 10.0 (66.06)
  NAPSI Score at Week 28 (n=9,7,44,38) | 34.9 (42.17) | 34.5 (44.21) | 52.0 (39.59) | 51.6 (49.97)
  NAPSI Score at Week 40 (n=9,7,42,36) | 31.6 (40.17) | 38.1 (48.80) | 59.9 (45.87) | 61.1 (53.17)
  NAPSI Score at Week 52 (n=9,7,42,37) | 48.0 (47.62) | 38.1 (48.80) | 60.0 (45.96) | 61.4 (48.28)
  NAPSI Score at Week 64 (n=9,7,42,36) | 51.5 (45.20) | 39.3 (45.32) | 56.6 (43.24) | 67.8 (37.49)

10. Secondary Outcome: Change From Baseline in the Number of Nails With Psoriasis Involvement at Week 12, 28, 40, 52 and 64
Description: The number of nails with psoriasis involvement was assessed by a dermatologist.
Time Frame: Week 12, 28, 40, 52 and 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Nails
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 16 | 64 | 61
Nails
  Change at Week 12 (n=15,16,62,61) | 0.9 (2.64) | -0.1 (0.25) | 0 (1.96) | 0 (1.83)
  Change at Week 28 (n=15,15,64,59) | -0.1 (2.80) | -0.1 (1.13) | -1.8 (2.89) | -1.4 (3.03)
  Change at Week 40 (n=15,15,61,56) | -1.5 (2.77) | -1.1 (3.20) | -2.6 (3.18) | -1.8 (3.34)
  Change at Week 52 (n=15,14,60,57) | -1.8 (3.23) | -1.4 (3.34) | -2.8 (3.32) | -1.92 (3.36)
  Change at Week 64 (n=15,14,60,56) | -1.3 (2.92) | -1.1 (3.32) | -2.6 (3.38) | -1.8 (3.43)

11. Secondary Outcome: Change From Baseline in Joint Symptoms Expressed on a Visual Analogue Scale (VAS) at Week 12, 28, 40, 52 and 64
Description: Each participant will assess his/her pain associated with joint symptoms on each assessment day using a 100 mm VAS ranging from 0 mm (no pain) to 100 mm (the worst pain imaginable).
Time Frame: Week 12, 28, 40, 52 and 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 2 | 1 | 6 | 13
Unit on scale
  Change at Week 12 (n=2,1,6,13) | 0.5 (0.71) | 23.0 (NA) — Standard deviation was not estimable because number of participant analyzed for this time point is 1 | -38.5 (28.93) | -9.3 (18.23)
  Change at Week 28 (n=2,0,6,12) | -8.0 (11.31) | NA (NA) — No participant was found with joint symptoms for which pain assessment could be conducted for this treatment group | -30.0 (37.97) | -24.8 (27.17)
  Change at Week 40 (n=2,0,6,11) | -16.0 (22.63) | NA (NA) — No participant was found with joint symptoms for which pain assessment could be conducted for this treatment group | -29.3 (33.17) | -30.2 (25.0)
  Change at Week 52 (n=2,0,6,11) | -4.0 (5.66) | NA (NA) — No participant was found with joint symptoms for which pain assessment could be conducted for this treatment group | -35.0 (35.49) | -28.1 (26.55)
  Change at Week 64 (n=2,0,6,11) | -7.5 (10.61) | NA (NA) — No participant was found with joint symptoms for which pain assessment could be conducted for this treatment group | -35.3 (38.55) | -27.2 (28.38)

12. Secondary Outcome: Percentage of Participants With Cleared (0), Cleared or Minimal (0 or 1) and Mild (Less Than or Equal to 2) Physician's Global Assessment (PGA) Score at Week 12
Description: Percentage of participants with PGA score of cleared (0), cleared or minimal (0 or 1) and mild (less than or equal to 2) was reported. The PGA score is a numeric scale which is completed by the physician and is designed to evaluate the physician's overall assessment of the participant's psoriasis. Overall lesions will be graded for induration (I), erythema (E), and scaling (S) as: 0=cleared, 1=minimal, 2=mild, 3=moderate, 4=marked, and 5=severe. The sum of the 3 scores (I + E + S) will be divided by 3 to obtain a final PGA score ranging from 0 [best] to 5 [worst].
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP)
Number analyzed (Participants) | 31 | 64 | 62
Percentage of participants | 9.7 | 57.8 | 69.4
Statistical Analysis 1: Comparison: Ustekinumab 45 mg (CP) vs Ustekinumab 90 mg (CP); Test type: Superiority or Other; p < 0.0001, Fisher Exact — Fisher's exact test (using Holm's method)

13. Secondary Outcome: Percentage of Participants With Cleared (0), Cleared or Minimal (0 or 1) and Mild (Less Than or Equal to 2) Physician's Global Assessment (PGA) Score at Week 64
Description: as for outcome 12
Time Frame: Week 64
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Number analyzed (Participants) | 15 | 14 | 60 | 56
Percentage of participants
  PGA score= 0 (cleared) | 13.3 | 21.4 | 21.7 | 28.6
  PGA score= 0 or 1 (minimal) | 53.3 | 71.4 | 53.3 | 69.6
  PGA score= 0, 1 or 2 (mild) | 73.3 | 71.4 | 83.3 | 82.1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72
Description: Safety population included all randomized participants who received at least one dose of the study drug.
Arm/Group | Placebo (CP) | Ustekinumab 45 mg (CP) | Ustekinumab 90 mg (CP) | Placebo A (After CP) | Placebo B (After CP) | Ustekinumab 45 mg (After CP) | Ustekinumab 90 mg (After CP)
Serious Adverse Events (participants affected / at risk) | 2/32 | 0/64 | 3/62 | 1/15 | 1/13 | 5/64 | 4/62
Other Adverse Events (participants affected / at risk) | 20/32 | 42/64 | 36/62 | 14/15 | 13/13 | 61/64 | 60/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=32) | Ustekinumab 45 mg (CP) (N=64) | Ustekinumab 90 mg (CP) (N=62) | Placebo A (After CP) (N=15) | Placebo B (After CP) (N=13) | Ustekinumab 45 mg (After CP) (N=64) | Ustekinumab 90 mg (After CP) (N=62)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=32) | Ustekinumab 45 mg (CP) (N=64) | Ustekinumab 90 mg (CP) (N=62) | Placebo A (After CP) (N=15) | Placebo B (After CP) (N=13) | Ustekinumab 45 mg (After CP) (N=64) | Ustekinumab 90 mg (After CP) (N=62)
Nasopharyngitis (Infections and infestations) | 3 | 10 | 10 | 8 | 9 | 35 | 29
Psoriasis (Skin and subcutaneous tissue disorders) | 7 | 1 | 2 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 7 | 0 | 2 | 2 | 13 | 8
Eosinophil count increased (Investigations) | 1 | 3 | 4 | 0 | 0 | 4 | 5
Liver function test abnormal (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 7
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 6
Folliculitis (Infections and infestations) | 0 | 1 | 2 | 2 | 0 | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infected epidermal cyst (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 3 | 8 | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 5 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 0 | 4 | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal atrophy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 11 | 12
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 2 | 3 | 6
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 5 | 4
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 5 | 3
Glucose urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 3 | 3
Lymphocyte count decreased (Investigations) | 0 | 3 | 0 | 1 | 0 | 5 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 3 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 4 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 3
Blood amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood cholesterol decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 5
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Basophil count increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on Principle investigator is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.